CLINICAL TRIAL: NCT05737576
Title: A Single Center, Randomized, Double-Blind, 2-period, 2-sequence Crossover Designed Study to Evaluate the Pharmacokinetics and Pharmacodynamics Between HR011408 and NovoRapid® in Healthy Subject
Brief Title: The Pharmacokinetics and Pharmacodynamics Between HR011408 and NovoRapid® in Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HR011408-102
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Intervention Model Description: Crossover Assigned to HR011408 or NovoRapid®
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): HR011408 injection + NovoRapid®
  Interventions: Drug: HR011408 injection; NovoRapid®
- Cohort 2 (Experimental): NovoRapid® + HR011408 injection
  Interventions: Drug: NovoRapid®；HR011408 injection
- Cohort 3 (Experimental): HR011408 injection + NovoRapid®
  Interventions: Drug: HR011408 injection; NovoRapid®
- Cohort 4 (Experimental): NovoRapid® + HR011408 injection
  Interventions: Drug: NovoRapid®；HR011408 injection
- Cohort 5 (Experimental)
  Interventions: Drug: HR011408 injection; NovoRapid®
- Cohort 6 (Experimental)
  Interventions: Drug: HR011408 injection; NovoRapid®

INTERVENTIONS:
Drug: HR011408 injection; NovoRapid® — HR011408 injection, administered subcutaneously in dose 1. NovoRapid®, administered subcutaneously in dose 1.
  Arms: Cohort 1
Drug: NovoRapid®；HR011408 injection — NovoRapid®, administered subcutaneously in dose 1. HR011408 injection, administered subcutaneously in dose 1.
  Arms: Cohort 2
Drug: HR011408 injection; NovoRapid® — HR011408 injection, administered subcutaneously in dose 2. NovoRapid®, administered subcutaneously in dose 2.
  Arms: Cohort 3
Drug: NovoRapid®；HR011408 injection — NovoRapid®, administered subcutaneously in dose 2. HR011408 injection, administered subcutaneously in dose 2.
  Arms: Cohort 4
Drug: HR011408 injection; NovoRapid® — HR011408 injection, administered subcutaneously in dose 3. NovoRapid®, administered subcutaneously in dose 3.
  Arms: Cohort 5
Drug: HR011408 injection; NovoRapid® — NovoRapid®, administered subcutaneously in dose 3. HR011408 injection, administered subcutaneously in dose 3.
  Arms: Cohort 6

SUMMARY:
The objective of the study is to compare the pharmacokinetics and pharmacodynamics between HR011408 and NovoRapid® in healthy subject.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained prior to any trial-related activities；
2. Male or female subjects aged 18-55 years (both inclusive) at the time of signing informed consent；
3. Body weight ≥50.0 kg for men and ≥45.0 kg for women, with body mass index (BMI) between 18.0 and 26.0 kg/m2 (both ends included)；
4. Are nonsmokers, have not smoked for at least 6 months before entering the study, and agree not to smoke (cigars, cigarettes, or pipes) or not use smokeless tobacco or nicotine products for the duration of the study.

Exclusion Criteria:

1. Have an abnormality in the 12-lead electrocardiogram (ECG) and as deemed to be clinically significant by the investigator;
2. have a significant history of the circulatory system, respiratory system, digestive system, urinary system, hematopoietic system, endocrine and metabolic system, neuropsychiatric system, musculoskeletal system, or existing diseases in the above systems may affect the safety of the subjects and interfere with the study data.
3. In the opinion of the investigator, are unsuitable for inclusion in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC0-0.5h) | from 0 to 30 minutes after dose administration
  Area under the concentration-time curve (AUC)

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC0-15min) | from 0 to 15 minutes after dose administration
Area under the concentration-time curve (AUC0-1h) | from 0 to 1 hour after dose administration
Area under the concentration-time curve (AUC0-1.5h) | from 0 to 1.5 hours after dose administration
Area under the concentration-time curve (AUC0-2h) | from 0 to 2 hours after dose administration
Area under the concentration-time curve (AUC0-10h) | from 0 to 10 hours after dose administration
Area under the concentration-time curve (AUC0-inf) | from 0 to infinity after dose administration
Onset of appearance | from 0 to 8 hours after dose administration
  First time point after dose administration when concentration reaches lower limit of quantification (LLOQ)
Time to 50% maximum observed concentration (time to 50% Cmax) | from 0 to 8 hours after dose administration
Time to maximum observed concentration (Tmax) | from 0 to 8 hours after dose administration
Maximum observed concentration (Cmax) | from 0 to 8 hours after dose administration
Elimination half-life (t1/2) | from 0 to 8 hours after dose administration
Area under the GIR-time curve (AUC) | from 0 to 10 hours after dose administration
  Area under the GIR-time curve (AUC0-10h)
Time to 50% maximum observed GIR(time to 50% GIRmax) | from 0 to 10 hours after dose administration
Time to maximum observed GIR (GIRmax) | from 0 to 10 hours after dose administration
Incidence and severity of adverse events (AEs) | from Day1 to Day14 after dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided